CLINICAL TRIAL: NCT06383000
Title: Assessment of the Effectiveness of the Continuous Non-invasive Haemodynamic Monitor
Brief Title: Assessment of Effectiveness of Continuous Non-invasive Haemodynamic Monitor by Compared to Invasive Blood Pressure and Pulse Oximeter Monitoring on Patients Undergoing General Anesthesia Surgeries for More Than 60 Minutes
Status: Not yet recruiting | Type: Observational
Sponsor: BLZ Technology (Wuhan) Co.,Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BLZ2024MOH
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: General Anesthesia; Blood Pressure; Pulse Rate; Arterial Line

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess whether the continuous non-invasive haemodynamic monitor MOH200 (measuring blood pressure as well as pulse rate) is effective or not in people undergoing general anesthetic surgeries for more than 60 minutes with planned invasive blood pressure and pulse oximeter monitoring.

Researchers will compare blood pressure data derived from MOH200 to the invasive blood pressure (IBP) data to see if the MOH200 is effective to measure the blood pressure of a surgical person. Also, researchers will compare pulse rate data drived from MOH200 to that from the pulse oximeter to see if the MOH200 is effective to measure the pulse rate of a surgical person.

Participants will be asked to be applied with MOH200 monitoring while IBP monitoring and pulse oximeter are applied. And after 30 minutes of the surgery, researchers will monitor the adverse effects occurred on the skin of participants to assess the safety of MOH200.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing general anesthesia surgeries for more than 60 minutes with IBP monitoring
2. Patients aging between 4 to 80 years old (including at least 5 pediatric subjects between 4 to 12 years old, and as for subjects over 12 years old, up to 60% of subjects between 12 to 50 years old, at least 15% of subjects between 50 to 60 years old, at least 15% of subjects between 60 to 70 years old, and at least 10% of subjects over 70 years old)
3. At least 30% of subjects is male and 30% is female
4. Volunteer to participate the study and sign the informed consent form willingly

Exclusion Criteria:

1. Patients with severe heart diseases which affect the stability of haemodynamics
2. Patients applied with the heart-lung machine, defibrillator or cardiopulmonary bypass
3. Patients with coagulation disorders, vasculopathy or vascular prostheses
4. Patients with cutaneous diseases, infections or trauma of the measured part of the body leading to failure of data acquisition
5. Patients with mental diseases, epilepsy or other diseases leading to involuntrary movements of the body
6. Patients with BMI no more than 17 or no less than 30 kg/m^2
7. Patients who are pregnant or at the unstable stage of diseases or with severe shock
8. Patients with infections or trauma at the position of artery cannulation, whose pulse is untouchable or who get positive in the Allen's test
9. Patients with diseases that the investigators think unsuitable for participating the study

Ages: 4 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients are going to undergoing a general anesthetic surgery for more than 60 minutes at the site (Tongji Hospital, Tongji Medical College of HUST) who are accord with the inclusion criteria and do not satisfy the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Continuous Non -invasive Blood Pressure Measurement from MOH200 | During the surgery
  The blood pressure is measured by MOH200 and recorded on the CRF for every 5 minutes, including mean blood pressure, diastolic blood pressure and systolic blood pressure.
Invasive Blood Pressure Measurement from Arterial Line | During the surgery
  The blood pressure is synchronously measured by the radial arterial line and also recorded on the CRF for every 5 minutes, including mean arterial pressure, diastolic blood pressure and systolic blood pressure.
Pulse Rate Measurement from MOH200 | During the surgery
  The pulse rate is measured by the MOH200 and recorded on the CRF for every 5 minutes.
Pulse Rate Measurement from Pulse Oximeter | During the surgery
  The pulse rate is measured by the pulse oximeter and recorded on the CRF for every 5 minutes during the surgery.

SECONDARY OUTCOMES:
The Occurrence of Pressure Pores | Once after all the subjects are recruited and the clinical trials are finished
  In order to evaluate the safety of the haemodynamic monitor MOH200, the occurrence of device-related pressure pores is recorded. The incidence of adverse reactions=(the number of pressure sore occurrence/the total number of subjects observed)×100%

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Zhou, Principal Investigator — Department of Anesthesiology, Tongji Hospital, Tongji Medical College of HUST

IPD SHARING:
Plan to Share IPD: No